CLINICAL TRIAL: NCT06855238
Title: Clinical Validation of an Artificial Intelligence Tool to Predict Inversion Time
Acronym: THAITI-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 09C335
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operator-set TI (control group) (No Intervention): During the cardiovascular magnetic resonance scan, the TI is set by an experienced human operator as per standard clinical practice
- THAITI-set TI (Experimental): During the cardiovascular magnetic resonance scan, the TI is set by the experimental software
  Interventions: Device: THAITI software

INTERVENTIONS:
Device: THAITI software — THAITI is an AI-based software which predicts on the fly personalised TI for late gadolinium enhancement imaging during cardiovascular magnetic resonance scans.
  The clinical investigators will be provided by the computer scientists investigators with a software, based on the developed AI model. During the CMR in the experimental group, investigators will input patients' data on the software (e.g. age, sex, dose of contrast…). The software will provide a TI value to be input in the MRI scanner. TI will be set accordingly to the AI prediction. A LGE series of 3 long axis (4-, 2- and 3-chambers view) and a short-axis stack will be acquired.
  For all the patients, a doctor expert in CMR will be at the scanner and quality check the images in real time. Every image where the myocardium is not optimally nulled will be repeated with a TI set by the CMR doctor.
  Arms: THAITI-set TI

SUMMARY:
Introduction: Inversion-recovery (IR) magnetic resonance (MR) sequences are commonly used to perform late-gadolinium enhancement (LGE) imaging during cardiac magnetic resonance (CMR) scans. Inversion Time (TI), i.e. the time between the 180° inverting pulse and the 90°-pulse, must be manually input to obtain optimal myocardium nulling. Determinants of this value are patient's, sequence, and contrast characteristics, and the time after contrast injection. The identification of the correct TI is pivotal to quality images. The determination of TI is mostly based on experience, and it can be challenging in some diseases and for less experienced operators.

Aim of this study is to test in a clinical setting an Artificial Intelligence (AI) tool, which we developed to automatically predict TI in CMR post-contrast IR LGE sequences, named "THAITI".

THAITI performance will be evaluated in terms of 1) quality of images obtained using the AI-predicted TI with a 4-point Likert scale; 2) quality of images obtained using the AI-predicted TI in terms of Contrast-Enhancement ratio, i.e. the signal intensity of enhanced/remote myocardium in CMR-LGE images; 3) numbers of images that need to be reacquired; 4) average time duration of CMR-LGE imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom CMR-LGE is performed for a clinical reason
* Mixed cardiac conditions (including cardiomyopathies, ischemic heart disease, normal scans, focal and diffuse myocardial pathological processes)
* Both sexes
* Any age
* Availability of serum creatinine, measured within one month prior to CMR
* Provision of the written informed consent

Exclusion Criteria:

* Non-contrast CMR
* First-pass perfusion stress-CMR
* Absolute contraindication to CMR
* Inadequate overall image quality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Images quality proportion | At examination
  Proportion of images with optimal/good quality

SECONDARY OUTCOMES:
contrast-enhancement ratio | At examination
  Contrast-Enhancement ratio (CER)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy